CLINICAL TRIAL: NCT00001100
Title: A Phase III Study to Evaluate the Safety and Efficacy of Ganciclovir (Dihydroxypropoxymethyl Guanine [DHPG]) Treatment of Symptomatic Central Nervous System (CNS) Congenital Cytomegalovirus (CMV) Infections.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMID ARB-AL-91-CMV; DAB-AL-558607
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Ganciclovir

INTERVENTIONS:
Drug: ganciclovir

SUMMARY:
The purpose of this study is to evaluate the benefits and safety of the antiviral drug ganciclovir (DHPG) given intravenously to treat newborn infants who are born infected with cytomegalovirus (CMV). CMV is a herpes virus that can infect most organs of the body, resulting in death in 10-30% of babies with symptoms of CMV. It can cause severe brain damage in a large percentage of surviving babies. Children in this study have a CMV infection of the central nervous system (CNS).

DETAILED DESCRIPTION:
The study will enroll 130 newborn infants 1 month of age or younger with CMV involving the CNS. Patients will be assigned randomly (like tossing a coin) to receive either DHPG or no study drug treatment. All babies in the study will receive standard of care treatment and clinical, diagnostic, laboratory, safety, and follow-up evaluations. Follow-up evaluations, including hearing and eye exams and developmental assessments, will be done periodically until the child reaches 5 years of age. The degree of improved hearing among surviving patients will be a primary measure of drug effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Infants may be eligible for this study if they:

* Were full term infants (at least 32 weeks gestation).
* Are 1 month of age or younger (preferably less than 2 weeks).
* Weighed at least 1,200 grams (2.5 lbs) at birth.
* Have confirmed cytomegalovirus.
* Have evidence of CMV infection of the CNS with or without evidence of other organ involvement.

Exclusion Criteria:

Infants will not be eligible for this study if they:

* Have concurrent bacterial infection.
* Have HIV infection.
* Have mild symptoms or no symptoms of CMV infection at birth.
* Have an abnormal brain development (hydranencephaly) or any devastating brain involvement.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130
Dates: Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- NIAID/DMID/CASG Central Unit, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Oliver SE, Cloud GA, Sanchez PJ, Demmler GJ, Dankner W, Shelton M, Jacobs RF, Vaudry W, Pass RF, Soong SJ, Whitley RJ, Kimberlin DW; National Institute of Allergy, Infectious Diseases Collaborative Antiviral Study Group. Neurodevelopmental outcomes following ganciclovir therapy in symptomatic congenital cytomegalovirus infections involving the central nervous system. J Clin Virol. 2009 Dec;46 Suppl 4(Suppl 4):S22-6. doi: 10.1016/j.jcv.2009.08.012. Epub 2009 Sep 18. PMID 19766534